CLINICAL TRIAL: NCT03398083
Title: A Human Abuse Potential Study to Evaluate the Subjective and Physiological Effects of Cannabidiol (CBD) Compared to Delta-9-Tetrahydrocannabinol (THC) and Alprazolam in an Inpatient Setting
Brief Title: Evaluation of the Effects of Cannabidiol (CBD) Compared to Delta-9-Tetrahydrocannabinol (THC) and Alprazolam
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Diagnostic
Other Study IDs: NIDA-CBD-Phase1-001
Record Dates: First submitted 2017-12-18; First posted 2018-01-12 (Actual); Last update posted 2018-06-14 (Actual); Status verified 2018-06

CONDITIONS: Cannabis Use Disorder
MeSH Terms: interventions — Dronabinol; Alprazolam

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (6):
- CBD (500 mg) (Active Comparator): CBD (500 mg) capsule by mouth one time during the 18 day treatment period
  Interventions: Drug: THC; Drug: Alprazolam; Drug: Placebo oral capsule
- CBD (1000 mg) (Active Comparator): CBD (1000 mg) capsule by mouth one time during the 18 day treatment period
  Interventions: Drug: THC; Drug: Alprazolam; Drug: Placebo oral capsule
- THC (2.5 mg) (Active Comparator): THC 2.5 mg capsule by mouth one time during the 18 day treatment period
  Interventions: Drug: Alprazolam; Drug: Placebo oral capsule; Drug: CBD
- THC (30 mg) (Active Comparator): THC 30 mg capsule by mouth one time during the 18 day treatment period
  Interventions: Drug: Alprazolam; Drug: Placebo oral capsule; Drug: CBD
- Alprazolam (Active Comparator): Alpraxolam 1.5 mg capsule by mouth one time during the 18 day treatment period
  Interventions: Drug: THC; Drug: Placebo oral capsule; Drug: CBD
- Placebo Oral Capsule (Placebo Comparator): Placebo capsule by mouth one time during the 18 day treatment period
  Interventions: Drug: THC; Drug: Alprazolam; Drug: CBD

INTERVENTIONS:
Drug: THC — THC capsule
  Arms: Alprazolam; CBD (1000 mg); CBD (500 mg); Placebo Oral Capsule
Drug: Alprazolam — Alpraxolam capsule
  Other Names: Xanax
  Arms: CBD (1000 mg); CBD (500 mg); Placebo Oral Capsule; THC (2.5 mg); THC (30 mg)
Drug: Placebo oral capsule — Sugar pill capsule
  Other Names: Placebo
  Arms: Alprazolam; CBD (1000 mg); CBD (500 mg); THC (2.5 mg); THC (30 mg)
Drug: CBD — CBD capsule
  Arms: Alprazolam; Placebo Oral Capsule; THC (2.5 mg); THC (30 mg)

SUMMARY:
The purpose of this study is to evaluate the abuse potential of CBD to determine whether it should remain as a Schedule I drug under the Controlled Substances Act, or be recommended for decontrol.

DETAILED DESCRIPTION:
This is a single-dose, randomized, double-blind, placebo- and active-controlled crossover study that evaluates CBD in comparison with THC, alprazolam, and placebo in healthy recreational drug users.

ELIGIBILITY:
Inclusion Criteria:

* Must understand and provide written informed consent prior to the initiation of any protocol-specific procedures.
* Male or female subjects 18 to 55 years of age, inclusive.
* Body mass index (BMI) within the range of 19.0 to 30.0 kg/m2, inclusive, and a minimum weight of at least 50.0 kg.
* Healthy, as determined by no clinically significant medical history, physical examination,
* 12-lead ECG, vital signs or laboratory (including hematology, clinical chemistry biochemistry, urinalysis, and serology) findings at Screening, as judged by the investigator.
* Must be a recreational drug user, defined as meeting all of the following criteria:

  * ≥10 lifetime non-therapeutic experiences (i.e., for psychoactive effects) with CNS depressants (e.g., benzodiazepines, barbiturates, zolpidem, eszopiclone, propofol/fospropofol, gamma-hydroxy-butyrate).
  * ≥10 lifetime non-therapeutic experiences with cannabinoids (e.g., cannabis, hashish, THC, nabilone).
  * At least 3 non-therapeutic uses of a sedative, and at least 3 non-therapeutic uses of a cannabinoid, within the 3 months prior to Screening.
* Must pass Qualification Phase eligibility criteria.
* Female subjects of childbearing potential who are not abstinent must be using and willing to continue using medically acceptable contraception throughout the trial and for 30 days after last dose. In the context of this trial, highly effective methods of contraception are defined as those, alone or in combination, that result in a low failure rate (i.e., less than 1% per year) when used consistently and correctly. Such methods include hormonal contraceptives, intrauterine devices/hormone-releasing systems, double-barrier methods, bilateral tubal occlusion, vasectomized partner, or sexual abstinence. Abstinence is only acceptable as true (total) abstinence, when this is in line with the preferred and usual lifestyle of the patient; periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception.
* Non-vasectomized male subjects must agree to a highly effective method of contraception with female partner(s) of childbearing potential and may not donate sperm throughout the trial and for 90 days after the last study drug administration.
* Able to speak, read, and understand English sufficiently to allow completion of all study assessments.
* Must be willing and able to abide by all study requirements and restrictions.

Exclusion Criteria:

* contact site directly for more information

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 42 (Actual)
Dates: Start 2017-12-04 (Actual); Primary Completion 2018-05-30 (Actual); Study Completion 2018-05-30 (Actual)

PRIMARY OUTCOMES:
Visual Analog Scale | 18 days
  Subjects will complete 13 scales. Each Visual Analog Scale is a self-administered assessment evaluating the subjective effects of a study agent. Subjects will be instructed to respond to the questions with regards to how they feel at that moment of the assessment on a 100 mm Likert Scale with 0 being "Not at all" and 100 being "Very" or "Extremely". All scales are unipolar or bipolar.

SECONDARY OUTCOMES:
Incidence of Increased Vital Signs | 25 days
  Number of participants with adverse events as assessed by vital signs
Incidence of Increased ECG Reading | 25 days
  Number of participants with adverse events as assessed by ECG
Incidence of Clinically Significant Laboratory Values | 25 days
  Number of participants with adverse events as assessed by laboratory changes

CONTACTS AND LOCATIONS:
Overall Officials: Debra Kelsh, MD, Principal Investigator — Vince and Associates Clinical Research
Locations (1):
- Debra Kelsh, MD, Overland Park, Kansas, United States